CLINICAL TRIAL: NCT00516399
Title: A Clinical Trial of the Treatment of Fungal Corneal Ulcers With Povidone-Iodine
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The DSMC decided it appeared futile to attempt to demonstrate non-inferiority of povidone-iodine to Natamycin.
Sponsor: University of California, Los Angeles (Other)
Collaborators: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Principal Investigator, Sherwin J. Isenberg, Chief, Division of Ophthalmology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 012488-01-00
Record Dates: First submitted 2007-08-14; First posted 2007-08-15 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Fungal Keratitis
Keywords: Fungal keratitis; povidone iodine; childhood blindness; povidone-iodine
MeSH Terms: interventions — Povidone-Iodine; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I: (Experimental): povidone-iodine 1.25% ophthalmic solution. The associated intervention descriptions contain sufficient information to describe the arm.
  Interventions: Drug: povidone-iodine 1.25% ophthalmic solution
- II (Active Comparator): natamycin ophthalmic suspension, USP 5%. The associated intervention descriptions contain sufficient information to describe the arm.
  Interventions: Drug: natamycin ophthalmic suspension, USP 5%

INTERVENTIONS:
Drug: povidone-iodine 1.25% ophthalmic solution
  Other Names: Betadine, Purdue Frederick, Norwalk
  Arms: I:
Drug: natamycin ophthalmic suspension, USP 5%
  Other Names: Natamet, M.J. Pharmaceuticals Ltd., Mumbai, India
  Arms: II

SUMMARY:
The purpose of this study is to determine the effectiveness of 1.25% povidone-iodine ophthalmic solution for the treatment of small to medium sized fungal corneal ulcers compared with an antifungal antibiotic.

DETAILED DESCRIPTION:
The medication to be studied is 1.25% povidone-iodine solution and the control medication is 5% natamycin ophthalmic suspension. The povidone-iodine concentration of 1.25% was chosen based on a study using povidone-iodine ophthalmic solution for the first week after ocular surgery. Initially, some patients complained of a stinging sensation when using the 2.5% concentration. This might prevent full compliance from some subjects. When the solution was diluted to 1.25%, there were no more complaints of discomfort. Therefore, in the actual one-week postoperative clinical trial, the 1.25 % concentration was used without any patient complaints and it was found to be effective. In a pilot study conducted in the Philippines, investigating treatment of small to medium-sized fungal corneal ulcers, 1.25% povidone-iodine was shown to be effective against fungal corneal ulcers including those caused by Fusarium solani and Mycelia sterila when treated for 7-20 days.

The povidone-iodine 1.25% solution will be prepared by removing 1.875 ml. of solution from a 15 ml. bottle of Balanced Salt Solution (BSS), (Alcon Laboratories, Inc., Fort Worth) and inserting 1.875 ml. of a 10% povidone-iodine solution (Betadine solution, Purdue Frederick, Norwalk). Preparations will be made weekly for each subject using sterile technique and are to be stored in a cool dark place. The control anti-fungal will be natamycin ophthalmic suspension, USP 5% (Natamet, M.J. Pharmaceuticals Ltd., Mumbai, India), which represents the current standard of care. The subjects will be discharged home on the same randomized medication that they were assigned while hospitalized.

Prospective candidates for the study, and/or their parent or guardian, will review the appropriate Human Subjects Consent Form, approved by the Human Subjects Protection Committee of the Harbor-UCLA Medical Center. After written consents, Informed and HIPPA, are obtained, each subject will be randomized to receive either povidone-iodine or the control drug. All subjects will be hospitalized for a minimum duration of 7 days for careful monitoring and appropriate treatment. To assure compliance, all these inpatient subjects will have their medications administered by medical personnel. Upon admission, the intake clinical examination will be recorded.

Each infected eye will be randomly assigned by the research nurse to be treated with povidone-iodine 1.25% or the control, anti-fungal medication natamycin. Randomization will be achieved by using random number generated randomization schedules. To guarantee similar distribution will occur, and not be left to chance, each study site randomization schedule will be stratified on ulcer sizes < 3mm. and > 3mm.

The only eye medications permitted beside povidone-iodine 1.25% ophthalmic solution and the control drug natamycin, will be atropine ophthalmic solution to reduce intraocular inflammation and prevent synechiae, and anti-glaucoma medication as needed. The atropine will be administered to the affected eye(s) twice a day and strength will vary according to the subject's age. Subjects less than 1 year of age will be given atropine 0.25%, ages 1-3 will be given 0.5%, and subjects greater than 3 years of age will be given 1%.

The dosing schedule of povidone-iodine 1.25% or control medication is as follows:

1. For the first three days, one drop of the medication will be applied every hour.
2. Day 4 and thereafter, hourly while awake, when asleep, every three hours. Sleep is not to exceed 9 hours. Treat all cases with intense drop therapy for a minimum of 5 days unless criteria for change in therapy are met.
3. At 5 days, decrease dosing frequency to every 2 hours while awake until "cured", only if no deterioration in any factor and improved in at least one factor, other than epithelial defect, is noted on 2 consecutive examinations.
4. If at 10 days the status remains unchanged, the subject is to exit the study.
5. After discharge, dosing frequency is to remain every 2 hours while awake until cured.

ELIGIBILITY:
Inclusion Criteria:

1. Be more than 1 month old.
2. Have a history of culture positive fungal corneal ulcer, that began within 14 days of presentation to the study center characterized by either a stromal defect with infiltrate or exudate, or a positive fungal stain on smear. Other clinical criteria to suspect fungal ulcers include firm (sometimes dry) elevated slough, "hyphate" lines extending beyond the ulcer edge into normal cornea, endothelial plaque, history of organic material striking the eye, intense inflammation of the cornea and anterior chamber, immune ring, Descemet's folds, multifocal granular (or feathery) grey-white satellite stromal infiltrates. A hypopyon may be present. The diameter of the ulcer will be between 1 mm and 6 mm, as long as there is no scleral involvement.
3. It is acceptable to enroll a subject who has received a graft, provided the graft meets the following requirements:

   1. The central ulcer is well within the donor cornea.
   2. There is no suture abscess.
   3. The graft has not previously failed.
4. The subject should not have a foreign body present on or in the cornea or eye. A subject can be enrolled after the foreign body is totally removed and the other enrollment criteria are met.

Exclusion Criteria:

1. The initial culture fails to show the presence of fungi.
2. The patient has a history of allergy to povidone-iodine, iodine, or natamycin.
3. The cornea or sclera has been perforated or perforation is impending.
4. The unaffected eye is legally blind.
5. Dacrocystitis is present.
6. Neurotrophic keratitis, exposure keratitis or keratitis sicca is present.
7. Prescribed topical or systemic steroids or other immunosuppressants are being used, unless discontinued before randomization.
8. The patient is known to be HIV positive.
9. The infiltrate extends into the posterior one-third of the stroma.
10. The initial culture shows significant growth of bacteria (>10 colonies).
11. Any topical antifungal agent has been used within the past week.
12. Both eyes are infected.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2008-03; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Number of days until disappearance of hypopyon and criteria for recovery and cure are met and subject is discharged home. Number of treatment failures. Ocular complications from the infection and ocular and systemic complications from the treatment. | Inferior outcome is defined as cure time under povidone-iodine treatment, which is at least 4 days longer than cure time under natamycin, or time until criteria for improvement to hospital discharge is reached.

CONTACTS AND LOCATIONS:
Overall Officials: Sherwin J. Isenberg, M.D., Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center